CLINICAL TRIAL: NCT06708221
Title: Real-Time IGRT: a Master Trial Assessing the Technical Feasibility of First-In-Human Real-Time Image Guided Radiation Therapy Methods
Brief Title: A Master Trial Assessing the Technical Feasibility of First-In-Human Real-Time Image Guided Radiation Therapy Methods
Acronym: Real-Time IGRT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sydney (Other)
Collaborators: Medical Research Future Fund (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RealTimeIGRT
Record Dates: First submitted 2024-11-13; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Cancer
Keywords: cancer; IGRT; radiotherapy; radiation therapy; Image Guided Radiation Therapy; breast cancer; lung cancer; Australia
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Real-Time IGRT (Experimental): Real-Time IGRT
  Interventions: Device: Real-Time Image Guided Radio Therapy (IGRT)

INTERVENTIONS:
Device: Real-Time Image Guided Radio Therapy (IGRT) — Real-time image guided radiation therapy (IGRT) methods image the cancerous tumour in real-time, enabling the treatment beam to focus its destructive energy on the patient's cancer, not their healthy tissue.

SUMMARY:
The goal of this clinical trial is to determine whether Real-Time Image Guided Radiation Therapy is a feasible method for radiation therapy delivery for patients with cancer.

The main questions it aims to answer are:

* Can all fractions per patient which are intended to be delivered with the real-time IGRT method be completed as planned?
* Can the beam accurately hit the tumour in ≥85% of fractions?
* Are there any unexpected grade >3 acute toxicities?

Participants will not require any additional treatments or preparation procedures above those required for normal radiation therapy treatment, to participate in this study.

DETAILED DESCRIPTION:
Real-time IGRT is a master trial to assess the technical feasibility of first-in-human real-time image guided radiation therapy methods.

Real-time image guided radiation therapy (IGRT) methods image the cancerous tumour in real-time, enabling the treatment beam to focus its destructive energy on the patient's cancer, not their healthy tissue. Using a real-time IGRT method available on scarce $10M MRI-guided radiation therapy devices, has halved the incidence of acute grade 2 or greater genitourinary (GU) toxicity for prostate cancer patients. However, >95% of radiotherapy is given on standard $3M devices. The halving in GU toxicity was confirmed in a study from Memorial Sloan-Kettering using combined kilovoltage and megavoltage guidance. This clinical benefit has led to a global demand: over 70% of centres want better real-time IGRT methods but are limited by resources and capacity. The tipping point is the implementation of real-time IGRT methods on standard devices. The Real-time IGRT trial addresses this unmet need by assessing an array of real-time IGRT methods.

To establish real-time IGRT methods, the University of Sydney partner hospitals and cancer centres have been working together across many different cancers, to create a database of images that have been, and are being, used to develop real-time IGRT methods. This development has led to the creation of LEARN, the Learning Environment for Artificial Intelligence in Radiotherapy New Technology, and the associated image acquisition study (https://clinicaltrials.gov/study/NCT05184790). The LEARN study looks at images retrospectively, meaning patients do not directly benefit from their involvement. To achieve benefit for study patients, and ultimately in broader practice, prospective implementation of real-time IGRT methods is required. This umbrella protocol, Real-time IGRT, enables a framework for the safe implementation and evaluation of real-time IGRT methods. Patient dosimetric and geometric targeting benefits will be measured, with the information acquired used to further improve the safety and accuracy of real-time IGRT methods.

The technologies being developed are numerous, covering different individual and combinations of imaging methods (surface, kV, MV), are applicable to different cancer sites, use marker and markerless approaches, and track one or more targets and normal tissues. To perform a feasibility study for each single innovation and for each single tumour site is time consuming when using a standard trial protocol. Instead, a master protocol trial comprises one general protocol that includes multiple subgroups and/or multiple interventions. Given this large variety of methods to be tested, a master protocol trial is the most efficient to maximise the safe testing of technologies, and to cease or pause technologies that do not meet the clinical requirements.

The master protocol trial aims to increase efficiency in terms of trial infrastructure and protocol administration to accelerate development of technical innovations in radiation oncology, meaning that patients benefit from the technologies earlier. By including multiple parallel cohorts, the protocol will accelerate the technical development of real-time IGRT methods and the evidenced-based introduction of real-time IGRT methods into clinical practice. This approach reduces the burden on the HREC, the sponsor and the participating centres.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older to be treated with curative radiation therapy
* Patients with brain, breast, head and neck, kidney, liver, lung, pancreas, prostate or spine cancer
* ECOG performance status 0-2
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Pregnancy,
* Patients with any other clinically significant medical condition which, in the opinion of the treating physician, makes it undesirable for the patient to participate in the study or which could jeopardize compliance with study requirements or severe psychiatric illness/social situation
* Additional inclusion and exclusion criteria may apply to a specific sub-study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Successful application of Real-Time IGRT | From the date of enrolment until 90 days after the completion of radiotherapy treatment
  Each real-time IGRT method under study is deemed feasible if successfully applied in 18 out of 20 consecutive patients (success rate of 90%), with a maximum of 40 patients to be included per cohort. If the real-time IGRT method is unsuccessfully applied in three consecutive patients or the real-time IGRT method is not successfully applied in 18 out of 20 consecutive patients after the inclusion of 40 patients, it is considered unfeasible. For each real-time IGRT method, success is defined by three general criteria (each of the three criteria should be met to reach feasibility):
  1. All fractions per patient which are intended to be delivered with the real-time IGRT method are completed as planned
  2. Absence of geographical miss in ≥85% of fractions or, in case of stereotactic treatments, in all minus one fraction. Geographical miss is defined as the clinical treatment volume outside the treated volume as measured on post-treatment image analysis
  3. No unexpected grade >3 acute toxicities

CONTACTS AND LOCATIONS:
Overall Officials: Paul Keall, Principal Investigator — University of Sydney
Locations (1):
- Liverpool Hospital, Liverpool, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Aligned with the NHMRC's Open Access Policy and the Health Studies Australian National Data Asset (HeSANDA) program, the Real-Time IGRT trial will aim to make the de-identified trial data publicly available for other scientific research via an external research data repository, archive or register. E.g. The Cancer Imaging Archives (TCIA, https://www.cancerimagingarchive.net/). Study data that are provided to an external research data repository will be stored at and managed by the external repository. Data will only be shared with repositories whose function has been reviewed and approved by an accredited Research Integrity/Ethics Committee/Board, under a Materials Transfer Agreement with the University.
Supporting Information: Study Protocol
Time Frame: Available following publication of final analysis, for a minimum of 5 years
Access Criteria: Researchers will be able to access de-identified trial information from an external research data repository, archive or register.